CLINICAL TRIAL: NCT03781726
Title: A Multi-Center, Open-Label Study of Glecaprevir/Pibrentasvir to Treat Recipients of Transplanted Kidneys From Deceased Donors With Hepatitis C Virus
Brief Title: Multi-center Study to Transplant Hepatitis-C Infected Kidneys
Acronym: MYTHIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Raymond Chung (Other)
Collaborators: AbbVie (Industry); University of Pennsylvania (Other); Johns Hopkins University (Other); University of Cincinnati (Other); Weill Medical College of Cornell University (Other); University of Michigan (Other); Northwestern University (Other)
Responsible Party: Sponsor-Investigator, Raymond Chung, Director of Hepatology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018P003140
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Renal Failure Chronic; Hepatitis C
Keywords: hemodialysis; renal failure; kidney transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hepatitis C; Renal Insufficiency | interventions — glecaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with glecaprevir/pibrentasvir Fixed Dose Combination (Experimental): 8 weeks of HCV treatment with combination tablet of glecaprevir and pibrentasvir
  Interventions: Drug: glecaprevir/pibrentasvir treatment

INTERVENTIONS:
Drug: glecaprevir/pibrentasvir treatment — combination treatment with glecaprevir and pibrentasvir fixed dose tablet.
  Other Names: Mavyret treatment

SUMMARY:
Open label multi center study for the donation of HCV positive kidneys to HCV negative recipients with interventional treatment to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
The study objective is to determine if the administration of the direct acting antiviral glecaprevir/pibrentasvir for 8 weeks after kidney transplantation is both safe and effective at preventing the spread of HCV infection from donor kidney with known HCV infection (all genotypes) to an HCV negative recipient as evidenced by a negative HCV viral RNA at 12 weeks post treatment.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Estimated glomerular filtration rate(eGFR) < 15 ml/min/1.73 m2
* Listed for an isolated kidney transplantation
* Able to understand and adhere to the study visit schedule and all other protocol requirements, and must voluntarily sign and date an informed consent
* No available medically acceptable, compatible living kidney donor
* Subject must agree to use an effective method of birth control per protocol specifications

Recipient Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to immunosuppressants utilized in kidney transplant
* Female who is pregnant, breastfeeding, or is planning to become pregnant during the course of the study
* History of HIV
* HCV RNA positive
* HBV surface Ag-positive or detectable HBV DNA
* Primary focal segmental glomerulosclerosis (FSGS) or disease process with increased risk of causing early graft failure as assessed by the transplant nephrologist and/or investigator team
* Presence of clinically significant liver disease
* Transplant candidate requiring antibody desensitization protocol for transplantation
* Most recent calculated panel reactive antibody (cPRA) >80%.
* Prior recipient of a non-renal solid organ transplant

Donor Organ Inclusion Criteria

* Deceased donor organ with kidney donor profile index (KDPI) ≤0.85
* HCV RNA-positive

Donor Organ Exclusion Criteria

* Known prior HCV treatment with direct acting antiviral medication
* HIV RNA-positive
* HBV Surface antigen-positive or HBV DNA-positive

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - Northwestern Medicine, Chicago, Illinois
  - John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Coded data is anticipated to be shared with collaborators in this multi-center consortium
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Real time
Access Criteria: researchers accessing IPD must be an approved site within the consortium.

REFERENCES:
- [Derived] Sise ME, Goldberg DS, Schaubel DE, Fontana RJ, Kort JJ, Alloway RR, Durand CM, Blumberg EA, Woodle ES, Sherman KE, Brown RS Jr, Friedewald JJ, Desai NM, Sultan ST, Levitsky J, Lee MD, Strohbehn IA, Landis JR, Fernando M, Gustafson JL, Chung RT, Reese PP. One-Year Outcomes of the Multi-Center StudY to Transplant Hepatitis C-InfeCted kidneys (MYTHIC) Trial. Kidney Int Rep. 2021 Dec 1;7(2):241-250. doi: 10.1016/j.ekir.2021.11.022. eCollection 2022 Feb. PMID 35155863

RESULTS

PARTICIPANT FLOW:
Groups:
- NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1): 8 weeks of HCV treatment with combination tablet of glecaprevir and pibrentasvir
  glecaprevir/pibrentasvir treatment: combination treatment with glecaprevir and pibrentasvir fixed dose tablet.
Period: Overall Study
Arm/Group | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1)
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1)
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [51 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Kidney disease etiology [Count of Participants; unit: Participants]
  Diabetic nephropathy | 11
  Hypertension | 9
  Polycystic kidney disease | 3
  Congenital/genetic | 2
  IgA nephropathy | 3
  Other | 2
On dialysis at baseline [Count of Participants; unit: Participants]
  Yes | 27
  No | 3
Time from consent to transplant [Median (Inter-Quartile Range); unit: Weeks] | 6.29 [1.86 to 10.1]
Time spent on waitlist at time of consent [Median (Inter-Quartile Range); unit: Weeks] | 137 [95 to 219]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Population: One patient missing BMI data
  kg/m^2
    number analyzed (Participants) | 29
    (all) | 29.5 [25.7 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable HCV
Description: HCV RNA < LLOQ 12 weeks after the last actual dose of G/P
Time Frame: 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1)
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Percentage of Subjects With On-treatment Virologic Failure
Description: HCV RNA > LLOQ during G/P treatment
Time Frame: During 8 week treatment course
Measure: Count of Participants; unit: Participants
Arm/Group | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1)
Number analyzed (Participants) | 30
Participants | 12

3. Secondary Outcome: Percentage of Subjects With Post-treatment Virologic Relapse
Description: HCV RNA > LLOQ after completion of G/P treatment and prior HCV RNA < LLOQ while on treatment
Time Frame: During 12 week post treatment follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1)
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline (day of transplant) to one year post transplant (1 year total)
Arm/Group | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1)
All-Cause Mortality (participants affected / at risk) | 2/30
Serious Adverse Events (participants affected / at risk) | 20/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1) (N=30)
neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) — not related to study drug/procedure
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — not related to study drug/procedure
postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) — not related to study drug/procedure
acute cellular rejection (Immune system disorders) | 2 (2) — not related to study drug/procedure
acute kidney injury (Renal and urinary disorders) | 1 (4) — not related to study drug/procedure
drug toxicity due to accidental overdosage (Injury, poisoning and procedural complications) | 1 (1) — not related to study drug/procedure
heart failure (Cardiac disorders) | 1 (1) — not related to study drug/procedure
stroke (Nervous system disorders) | 1 (1) — not related to study drug/procedure
vomiting (Gastrointestinal disorders) | 1 (1) — not related to study drug/procedure
hypotension (Respiratory, thoracic and mediastinal disorders) | 2 (2) — not related to study drug/procedure
gastritis (Gastrointestinal disorders) | 2 (3) — not related to study drug/procedure
hemorrhoidal hemorrhage (Blood and lymphatic system disorders) | 1 (1) — not related to study drug/procedure
small intestinal obstruction (Gastrointestinal disorders) | 1 (1) — not related to study drug/procedure
ileus (Gastrointestinal disorders) | 1 (2) — not related to study drug/procedure
renal calculi (Renal and urinary disorders) | 1 (1) — not related to study drug/procedure
abdominal infection (Gastrointestinal disorders) | 1 (3) — not related to study drug/procedure
coronavirus infection (Infections and infestations) | 1 (1) — not related to study drug/procedure
post procedural urine leak (Renal and urinary disorders) | 1 (1) — not related to study drug/procedure
fever (Infections and infestations) | 1 (1) — not related to study drug/procedure
renal graft function delayed (Renal and urinary disorders) | 1 (1) — not related to study drug/procedure
dysuria (Renal and urinary disorders) | 1 (1) — not related to study drug/procedure
cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) — not related to study drug/procedure
sepsis (Infections and infestations) | 1 (1) — not related to study drug/procedure
constipation (Gastrointestinal disorders) | 1 (1) — not related to study drug/procedure
syncope (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not related to study drug/procedure
chest pain (Cardiac disorders) | 1 (1) — not related to study drug/procedure
urinary tract obstruction (Renal and urinary disorders) | 1 (1) — not related to study drug/procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAT+ Kidney Transplant Treatment With Glecaprevir/Pibrentasvir Fixed Dose Combination (Arm 1) (N=30)
abdominal pain (Gastrointestinal disorders) | 6 (6) — not related to study drug/procedures
acute cellular rejection (Immune system disorders) | 2 (2) — not related to study drug/procedures
acute kidney injury (Renal and urinary disorders) | 2 (5) — not related to study drug/procedures
anemia (Blood and lymphatic system disorders) | 2 (2) — not related to study drug/procedures
anxiety (Psychiatric disorders) | 2 (2) — not related to study drug/procedures
bladder spasm (Renal and urinary disorders) | 2 (2) — not related to study drug/procedures
chills (General disorders) | 2 (2) — not related to study drug/procedures
constipation (Gastrointestinal disorders) | 2 (2) — not related to study drug/procedures
creatinine increased (Renal and urinary disorders) | 3 (3) — not related to study drug/procedures
cytomegalovirus infection reactivation (Infections and infestations) | 2 (2) — not related to study drug/procedures
dizziness (Nervous system disorders) | 7 (8) — not related to study drug/procedures
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) — not related to study drug/procedures
edema limbs (Vascular disorders) | 3 (3) — not related to study drug/procedures
fatigue (General disorders) | 3 (3)
gastritis (Gastrointestinal disorders) | 3 (3) — not related to study drug/procedures
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) — not related to study drug/procedures
headache (Nervous system disorders) | 3 (3) — not related to study drug/procedures
hyperglycemia (Endocrine disorders) | 6 (6) — not related to study drug/procedures
hyperkalemia (Renal and urinary disorders) | 4 (5) — not related to study drug/procedures
hypertension (Vascular disorders) | 5 (5) — not related to study drug/procedures
hypotension (Vascular disorders) | 5 (6) — not related to study drug/procedures
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — not related to study drug/procedures
nausea (General disorders) | 3 (3)
neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) — not related to study drug/procedures
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — not related to study drug/procedures
platelet count decreased (Blood and lymphatic system disorders) | 2 (2) — not related to study drug/procedures
renal graft function delayed (Renal and urinary disorders) | 2 (2) — not related to study drug/procedures
tremor (Nervous system disorders) | 5 (5) — not related to study drug/procedures
urinary retention (Renal and urinary disorders) | 3 (3) — not related to study drug/procedures
urinary tract infection (Renal and urinary disorders) | 3 (7) — not related to study drug/procedures
vomiting (Gastrointestinal disorders) | 3 (3) — not related to study drug/procedures
white blood cell count decreased (Blood and lymphatic system disorders) | 4 (5) — not related to study drug/procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT03781726/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT03781726/SAP_001.pdf